CLINICAL TRIAL: NCT00143091
Title: A Six-Week, Fixed Dose, Double-Blind, Double-Dummy, Placebo and Sertraline Controlled, Multicentre Trial to Evaluate the Safety and Efficacy of CP-316,311 in Outpatients With Major Depressive Disorder
Brief Title: Multicentre Trial to Evaluate the Safety and Efficacy of CP-316,311 in Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2211002
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder, Recurrent
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CP-316,311
Drug: Placebo
Drug: Sertraline

SUMMARY:
A six week, fixed dose, double-blind, double-dummy, placebo, and active controlled, multicentre trial to evaluate the safety and efficacy of CP-316,311 in outpatients with major depressive disorder.

DETAILED DESCRIPTION:
This study was terminated on March 17th, 2006. The results of the primary analysis at the interim showed that the CP-316,311 group was not significantly different than the placebo on the primary endpoint and therefore the data monitoring committee recommended termination of the trial. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with DSM-IV major depressive disorder

Exclusion Criteria:

* Women of child bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-04; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HAM-D (17) at the week 6 visit

SECONDARY OUTCOMES:
Change from baseline in MADRS, HAM-A, CGI-S and CGI-I at the week 6 visit.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (2):
  - Pfizer Investigational Site, Bellevue, Washington
  - Pfizer Investigational Site, Seattle, Washington
- Russia (4):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Rostov-on-Don
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Smolensk
- Serbia and Montenegro (4):
  - Pfizer Investigational Site, Belgrade, Serbia
  - Pfizer Investigational Site, Kragujevac, Serbia
  - Pfizer Investigational Site, Novi Sad, Serbia
  - Pfizer Investigational Site, Belgrade

REFERENCES:
- [Derived] Binneman B, Feltner D, Kolluri S, Shi Y, Qiu R, Stiger T. A 6-week randomized, placebo-controlled trial of CP-316,311 (a selective CRH1 antagonist) in the treatment of major depression. Am J Psychiatry. 2008 May;165(5):617-20. doi: 10.1176/appi.ajp.2008.07071199. Epub 2008 Apr 15. PMID 18413705
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2211002&StudyName=Multicentre+Trial+to+Evaluate+the+Safety+and+Efficacy+of+CP%2D316%2C311+in+Major+Depressive+Disorder+